CLINICAL TRIAL: NCT06395259
Title: Evaluation of the Oxidative Status of Patients Undergoing Solid Organs Transplantation: Observational Study
Brief Title: Observational Study on the Variation of Ascorbic Acid in Patients Undergoing Solid Organ Transplantation
Acronym: REDOX-TX
Status: Active, not recruiting | Type: Observational
Sponsor: Policlinico Hospital (Other)
Responsible Party: Principal Investigator, Giacomo Grasselli, MD, University of Milan
Other Study IDs: 3334
Record Dates: First submitted 2024-01-24; First posted 2024-05-02 (Actual); Last update posted 2024-09-04 (Actual); Status verified 2024-09

CONDITIONS: Transplantation; Ascorbic Acid Deficiency
Keywords: Transplantation; Ascorbic Acid; Oxidative Stress; Primary Graft Dysfunction
MeSH Terms: conditions — Ascorbic Acid Deficiency; Primary Graft Dysfunction

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Whole blood samples are collected (in lithium-heparin tubes), appropriately centrifuged, and the plasma thus obtained is frozen at -80°
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Hypovitaminosis Group: Patients who at the end of surgery have sub-optimal plasma ascorbic acid levels, i.e. with concentrations lower than 28 µmol/L
- Normal Range Group: Patients who at the end of surgery have plasma ascorbic acid levels equal to or greater than 28 µmol/L

SUMMARY:
The objective of this observational clinical study is to evaluate the variations in ascorbic acid during the transplantation phases and how these variations influence the oxidative status and patient outcome.

The main questions it aims to answer are:

* how many patients arrive at the transplant in a state of hypovitaminosis C?
* how does hypovitaminosis C affect the patient's oxidative status?
* how does hypovitaminosis C affect the length of stay in intensive care and post-transplant complications?

DETAILED DESCRIPTION:
Researches will compared:

Differences between Hypovitaminosis Group and Normal Range Group Changes in oxidative stress markers before and after solid organ transplantation Incidence of allograft dysfunction between groups Incidence of acute kidney injury and other complications between groups

ELIGIBILITY:
Inclusion Criteria:

* Adult patients undergoing solid organ transplantation (liver or kidney or lung)

Exclusion Criteria:

* Minor patients
* Multi-organ transplantation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing liver, lungs or kidneys transplantation at Ospedale Maggiore in Milan. There is no control group
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2024-08-31 (Actual); Study Completion 2024-08-31 (Estimated)

PRIMARY OUTCOMES:
Ascorbic Acid levels | At induction of anesthesia for TX, within 24h from ICU admission, 72 hours after transplantation, 7 days after transplantation
  Quantification of plasma ascorbic acid levels before and after liver/kidney/lung transplantation

SECONDARY OUTCOMES:
Reactive Oxygen Species (ROS) levels | At induction of anesthesia for TX, within 24 hours from ICU admission, 72 hours after transplantation, 7 days after transplantation
  Quantification of ROS before and after liver/kidney/lung transplantation
Total Antioxidant Capacity (TAC) levels | At induction of anesthesia for TX, within 24 hours from ICU admission, 72 hours after transplantation, 7 days after transplantation
  Quantification of TAC before and after liver/kidney/lung transplantation
8-hydroxydeoxyguanosine (8-OHdG) levels | At induction of anesthesia TX, within 24 hours from ICU admission, 72 hours after transplantation, 7 days after transplantation
  Quantification of 8-OHdG before and after liver/kidney/lung transplantation
Mechanical ventilation | From ICU admission until extubation occurs, assessed daily up to 100 days from transplantation
  Duration of mechanical ventilation (days) until extubation of the recipient
Length of Intensive Care Unit (ICU) stay | From ICU admission until ICU discharge occurs, assessed daily up to 100 days from transplantation
  Length of ICU stay
Allograft dysfunction | Within the first 7 days after transplantation
  Incidence of early allograft dysfunction (EAD in liver recipients), primary graft dysfunction (PGD in lung recipients), delayed graft function (DGF in kidney recipients)
Mortality in Intensive Care Unit (ICU) | From ICU admission until ICU discharge occurs, assessed daily up to 100 days from transplantation
  Incidence of death for any cause during ICU stay
Length of hospitalization | From ICU admission until hospital discharge occurs, assessed daily up to 100 days from transplantation
  Length of stay in hospital (days)
Acute kidney injury (AKI) | Worst kidney function within the first 7 days after TX
  Incidence of postoperative renal injury after liver/kidney/lung transplantation as Kidney Disease Improving Global Outcomes (KDIGO) criteria

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico di Milano, Milan, Italy

REFERENCES:
- [Background] Fernandez AR, Sanchez-Tarjuelo R, Cravedi P, Ochando J, Lopez-Hoyos M. Review: Ischemia Reperfusion Injury-A Translational Perspective in Organ Transplantation. Int J Mol Sci. 2020 Nov 13;21(22):8549. doi: 10.3390/ijms21228549. PMID 33202744
- [Background] Pak O, Sydykov A, Kosanovic D, Schermuly RT, Dietrich A, Schroder K, Brandes RP, Gudermann T, Sommer N, Weissmann N. Lung Ischaemia-Reperfusion Injury: The Role of Reactive Oxygen Species. Adv Exp Med Biol. 2017;967:195-225. doi: 10.1007/978-3-319-63245-2_12. PMID 29047088
- [Background] Shi S, Xue F. Current Antioxidant Treatments in Organ Transplantation. Oxid Med Cell Longev. 2016;2016:8678510. doi: 10.1155/2016/8678510. Epub 2016 Jun 15. PMID 27403232
- [Background] Williams A, Riise GC, Anderson BA, Kjellstrom C, Schersten H, Kelly FJ. Compromised antioxidant status and persistent oxidative stress in lung transplant recipients. Free Radic Res. 1999 May;30(5):383-93. doi: 10.1080/10715769900300421. PMID 10342331
- [Background] Kumar S, Sharma U, Sharma A, Kenwar DB, Singh S, Prasad R, Minz M. Evaluation of oxidant and antioxidant status in living donor renal allograft transplant recipients. Mol Cell Biochem. 2016 Feb;413(1-2):1-8. doi: 10.1007/s11010-015-2617-6. Epub 2016 Jan 13. PMID 26762627
- [Background] Sotomayor CG, Eisenga MF, Gomes Neto AW, Ozyilmaz A, Gans ROB, Jong WHA, Zelle DM, Berger SP, Gaillard CAJM, Navis GJ, Bakker SJ. Vitamin C Depletion and All-Cause Mortality in Renal Transplant Recipients. Nutrients. 2017 Jun 2;9(6):568. doi: 10.3390/nu9060568. PMID 28574431
- [Background] Hill A, Borgs C, Fitzner C, Stoppe C. Perioperative Vitamin C and E levels in Cardiac Surgery Patients and Their Clinical Significance. Nutrients. 2019 Sep 9;11(9):2157. doi: 10.3390/nu11092157. PMID 31505814
- [Background] Borran M, Dashti-Khavidaki S, Alamdari A, Naderi N. Vitamin C and kidney transplantation: Nutritional status, potential efficacy, safety, and interactions. Clin Nutr ESPEN. 2021 Feb;41:1-9. doi: 10.1016/j.clnesp.2020.12.017. Epub 2021 Jan 9. PMID 33487249
- [Background] Frei B, Stocker R, England L, Ames BN. Ascorbate: the most effective antioxidant in human blood plasma. Adv Exp Med Biol. 1990;264:155-63. doi: 10.1007/978-1-4684-5730-8_24. PMID 2244489
- [Background] Oudemans-van Straaten HM, Spoelstra-de Man AM, de Waard MC. Vitamin C revisited. Crit Care. 2014 Aug 6;18(4):460. doi: 10.1186/s13054-014-0460-x. PMID 25185110
- [Background] Spoelstra-de Man AME, Elbers PWG, Oudemans-van Straaten HM. Making sense of early high-dose intravenous vitamin C in ischemia/reperfusion injury. Crit Care. 2018 Mar 20;22(1):70. doi: 10.1186/s13054-018-1996-y. PMID 29558975
- [Background] Wang Y, Lin H, Lin BW, Lin JD. Effects of different ascorbic acid doses on the mortality of critically ill patients: a meta-analysis. Ann Intensive Care. 2019 May 20;9(1):58. doi: 10.1186/s13613-019-0532-9. PMID 31111241
- [Background] Gori F, Fumagalli J, Lonati C, Caccialanza R, Zanella A, Grasselli G. Ascorbic acid in solid organ transplantation: A literature review. Clin Nutr. 2022 Jun;41(6):1244-1255. doi: 10.1016/j.clnu.2022.04.004. Epub 2022 Apr 12. PMID 35504167